CLINICAL TRIAL: NCT05532176
Title: Determination of Standards on a New Static and Dynamic Posture Platform
Brief Title: Posture Standards of a New Dynamic Platform
Acronym: VESTINORM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00856-37
Record Dates: First submitted 2022-08-25; First posted 2022-09-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Static and Dynamic Posture Standards
Keywords: vertigo; posture; platform; diagnostic; physiotherapist; balance; standards; algorithm
MeSH Terms: conditions — Vertigo; Disease

STUDY DESIGN:
Intervention Model Description: seven sub-groups of 40 persons each according to their age: 20-29/30-39/40-49/50-59/60-69/70-79/80-89years old
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- postural group (Other): one healthy group of different age
  Interventions: Other: Posture standards

INTERVENTIONS:
Other: Posture standards — Dynamic and static Postural measurements according to four types of tests

SUMMARY:
The objective is the determination of norms on healthy subjects, by age groups (20-29/30-39/40-49/50-59/60-69/70-79/80-89 years) for the posturological evaluation of four posture tests: the sensory organization test, the motor coordination test, the adaptation test, the stability limit test.

DETAILED DESCRIPTION:
The objective is the determination of norms by age groups (20-29/30-39/40-49/50-59/60-69/70-79/80-89) of four tests of posture: the test of sensory organization, the test of motor coordination, the test of adaptation, the test of stability limit, of a new platform of static and dynamic posturology.

When moving within an environment, sensory information from the environment and the body is registered within the sensory systems (Hilber et al., 2018). More specifically, it is the functions of balancing and spatial orientation that are brought into play to produce behavioral responses that are adapted to different situations and to anticipate events in one's environment. It is therefore essential to establish not only posturological norms but also norms for the function of spatial orientation in order to propose a complete assessment of the postural and spatial cognitive profile of healthy subjects that can serve as a reference population.

These standards will serve as a basis for determining the pathological values during the exploration of numerous pathologies, in particular vestibular pathology, pathologies inducing balance and posture disorders (neurology, rheumatology).

The measurement of posture and variations of the center of gravity represents an important output marker, little or never taken into account in medical practice, and linked to a large number of integration processes, in particular multisensory and sensory-motor. Its parameters vary according to the sensory information received and processed related to the maintenance of balance: visual system, vestibular system, somesthesic system, visceral sensory system. Posture is also modulated by the attentional level and cognitive load. Posturography is one of the most cost-effective instruments in terms of clinical utility, particularly in the diagnosis of vestibular pathology (Stewart et al., 1999). Thus, the development of such an instrument represents an innovative and advantageous development in terms of diagnostic improvement.

the investigators will perform the standard setting according to a precise statistical approach (analysis of variance ANOVA with correlation coefficients and 95% confidence intervals to establish test-retest reliability).

ELIGIBILITY:
Inclusion Criteria:

* No symptoms of vertigo, dizziness, balance disorders, motion sickness;
* No history of neurological or musculoskeletal pathology;
* No history of neurological or musculoskeletal pathology; -No known medication or medication likely to modify balance;
* No history of two or more falls in the six months preceding the study;
* No psychiatric disorder;
* Normal vision with or without correction;
* Be able to stand for more than 20 minutes and walk independently

Exclusion Criteria:

* Subjects under 20 years of age
* Pregnant or breastfeeding women,
* Persons in an emergency situation or unable to give their consent, including adults under guardianship
* Persons under legal protection
* Persons deprived of liberty, minors, protected adults,
* Inclusion of the subject in another interventional research protocol with pharmacological objectives during the present study

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female sub-groups of 20 people each per group of age.
Enrollment: 260 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Sensory Organization Test (SOT) | day 1 after inclusion
  Standards (arbitrary unit)
Sensory Organization Test (SOT) | day 15 after inclusion
  Standards (arbitrary unit)
Motor Coordination Test (MCT) | day 1 after inclusion
  Standards (arbitrary unit)
Motor Coordination Test (MCT) | day 15 after inclusion
  Standards (arbitrary unit)
Adaptation Test (ADT) | day 1 after inclusion
  Standards (arbitrary unit)
Adaptation Test (ADT) | day 15 after inclusion
  Standards (arbitrary unit)
Limits of Stability Test (LOS) | day 1 after inclusion
  Standards (arbitrary unit)
Limits of Stability Test (LOS) | day 15 after inclusion
  Standards (arbitrary unit)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No